CLINICAL TRIAL: NCT01849640
Title: Active Surveillance for P. Falciparum Drug Resistance With Assessment of Transmission Blocking Activity of Single Dose Primaquine in Cambodia
Brief Title: Antimalarial Drug Resistance With Assessment of Transmission Blocking Activity
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor efficacy of DHA-piperaquine due to likely drug resistance.
Sponsor: David Saunders (Other Government)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Royal Cambodian Armed Forces (Unknown); US Department of Defense Armed Forces Health Surveillance Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Saunders, David Saunders, LTC, MC, USA, Armed Forces Research Institute of Medical Sciences, Thailand
Organization: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR#1877; HRPO Log Number A-17145 (Other: USAMRMC ORP HRPO)
Record Dates: First submitted 2013-02-27; First posted 2013-05-08 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Malaria; Drug resistance; DHA-piperaquine; Cambodia; Transmission Blocking
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA-piperaquine with Primaquine (Active Comparator): 3-day treatment course of DHA-piperaquine with 45mg single dose primaquine
  Interventions: Drug: DHA-piperaquine and Primaquine
- DHA-piperaquine without Primaquine (Active Comparator): 3-day treatment course of DHA-piperaquine
  Interventions: Drug: DHA-piperaquine and Primaquine

INTERVENTIONS:
Drug: DHA-piperaquine and Primaquine — Subject will be enrolled in open label fashion to a 3-day treatment course of DHA-piperaquine (DP) by directly observed therapy (DOT, all patients will receive a total of 9 tablets containing 40mg DHA and 320mg of piperaquine in divided doses at 0, 24 and 48 hours (3 tablets once per day) for the 3 day course. At completion of DP treatment volunteers will be randomized in an open label fashion to receive a single 45 mg dose of primaquine or no therapy.

SUMMARY:
This is a two-arm, open label Treatment Study comparing the efficacy, safety, tolerability and pharmacokinetics of a three-day course of Dihydroartemisinin-Piperaquine (DP) with or without single-dose primaquine in patients with uncomplicated Plasmodium falciparum malaria. On the last day of DP therapy, volunteers will be randomized to receive either a single 45 mg dose of primaquine (PQ) or DP treatment only (no primaquine).

DETAILED DESCRIPTION:
Volunteers with uncomplicated malaria in Cambodia will be enrolled to current standard of care therapy with DHA-piperaquine to monitor therapeutic efficacy and measure resistance. The cardiac safety of piperaquine will be monitored with electrocardiograms during the treatment period. Resistance to DP and DP-PQ will be assessed by a combination of clinical, pharmacologic, and parasitologic parameters including genomic signatures of selection during careful weekly follow-up visits for 42 days. Volunteers will be randomized on day 3 to either a single 45mg dose of primaquine or no sexual stage therapy to evaluate effects of primaquine on the sexual stages of malaria (gametocytes) and potential transmissibility of infection to Anopheles mosquitoes as compared to those not treated with primaquine.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer with uncomplicated P. falciparum malaria (volunteers with mixed P. falciparum and P. vivax infections may be enrolled), 18-65 years of age
2. Baseline asexual parasite density between 1,000-200,000 parasites/uL
3. Able to provide informed consent
4. Available and agree to follow-up for anticipated study duration including 3 day treatment course at the MTF and weekly follow-up for the 42-day period
5. Authorized by local commander to participate if active duty military

Exclusion Criteria:

1. Allergic reaction or contraindication to DHA, piperaquine or primaquine
2. Significant acute comorbidity requiring urgent medical intervention
3. Signs/symptoms and parasitological confirmation of severe malaria
4. Use of any anti-malarial within the past 14 days.
5. Class I or II G6PD deficiency (defined as severe) as determined at screening
6. Pregnant or lactating female, or female of childbearing age, up to 50 years of age, who does not agree to use an acceptable form of contraception during the study
7. Clinically significant abnormal EKG, including a QTcF interval > 500 ms at enrollment.
8. Known or suspected concomitant use of QTc prolonging medications.
9. Judged by the investigator to be otherwise unsuitable for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of DP | 3 years
  Efficacy rates at 42 days (with 95% confidence intervals) for DP with and without single dose primaquine for uncomplicated P. falciparum diagnosed by positive PCR-corrected malaria microscopy.

SECONDARY OUTCOMES:
Efficacy of Primaquine to treat sexual stage gametocyte infection and prevent transmission of P. falciparum gametocytes to mosquitoes. | 3 years
  To detect efficacy of a onetime dose of primaquine after completion of therapy for blood stage infection on gametocytemia that may persist after DP treatment by using comparative rates of sexual stage infections between patients dosed with and without primaquine based on a composite endpoint of light microscopy and PCR detection and staging of gamteocytes with mosquito membrane feeding assay to detect oocysts in sterile lab-reared mosquitoes.

CONTACTS AND LOCATIONS:
Overall Officials: David Saunders, MD, MPH, Principal Investigator — Dept. of Immunology and Medicine, Armed Forces Research Institute of Medical Sciences (AFRIMS)
Locations (1):
- Anlong Veng Referral Hospital, Anlong Veaeng, Oddormean Chey, Cambodia

REFERENCES:
- [Background] Saunders DL, Vanachayangkul P, Lon C; U.S. Army Military Malaria Research Program; National Center for Parasitology, Entomology, and Malaria Control (CNM); Royal Cambodian Armed Forces. Dihydroartemisinin-piperaquine failure in Cambodia. N Engl J Med. 2014 Jul 31;371(5):484-5. doi: 10.1056/NEJMc1403007. No abstract available. PMID 25075853
- [Result] Spring MD, Lin JT, Manning JE, Vanachayangkul P, Somethy S, Bun R, Se Y, Chann S, Ittiverakul M, Sia-ngam P, Kuntawunginn W, Arsanok M, Buathong N, Chaorattanakawee S, Gosi P, Ta-aksorn W, Chanarat N, Sundrakes S, Kong N, Heng TK, Nou S, Teja-isavadharm P, Pichyangkul S, Phann ST, Balasubramanian S, Juliano JJ, Meshnick SR, Chour CM, Prom S, Lanteri CA, Lon C, Saunders DL. Dihydroartemisinin-piperaquine failure associated with a triple mutant including kelch13 C580Y in Cambodia: an observational cohort study. Lancet Infect Dis. 2015 Jun;15(6):683-91. doi: 10.1016/S1473-3099(15)70049-6. Epub 2015 Apr 12. PMID 25877962
- [Derived] Vanachayangkul P, Lon C, Spring M, Sok S, Ta-Aksorn W, Kodchakorn C, Pann ST, Chann S, Ittiverakul M, Sriwichai S, Buathong N, Kuntawunginn W, So M, Youdaline T, Milner E, Wojnarski M, Lanteri C, Manning J, Prom S, Haigney M, Cantilena L, Saunders D. Piperaquine Population Pharmacokinetics and Cardiac Safety in Cambodia. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02000-16. doi: 10.1128/AAC.02000-16. Print 2017 May. PMID 28193647
- See also: Interim Results — http://www.nejm.org/doi/full/10.1056/NEJMc1403007